CLINICAL TRIAL: NCT00460616
Title: Observational Study to Investigate the Prevalence of Cardiac Abnormalities and Valvular Regurgitation in Patients With Prolactinomas Treated Chronically With Cabergoline
Brief Title: Cardiac Valve Complications in Prolactinomas Treated With Cabergoline
Acronym: ValveCab
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Department of Mol and Clin Endocrinol Oncol
Other Study IDs: NeuroendoUnit-2
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2007-10

CONDITIONS: Prolactinomas
Keywords: Prolactin; Prolactinomas; Dopamine-Agonists; Cabergoline; Cardiac valve disease
MeSH Terms: conditions — Prolactinoma; Heart Valve Diseases | interventions — Cabergoline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients already receiving treatment with cabergoline.
  Interventions: Drug: Cabergoline
- 2: healthy controls sex and age-matched with the patients

INTERVENTIONS:
Drug: Cabergoline — According with our previous studies, in the patients with microprolactinoma and in those with non-tumoral hyperprolactinemia, cabergoline treatment was administered orally at a starting dose of 0.25 mg twice weekly for the first two weeks and then 0.5 mg twice weekly. After 2 months of treatment, dose adjustment was carried out every 2 months on the basis of serum PRL suppression.
  Other Names: Dostinex
  Groups: 1

SUMMARY:
Dopamine agonists are first-line agents for the treatment of prolactinomas (1) and Parkinson's disease (2). There is evidence supporting a causal relationship between the occurrence of drug-induced "restrictive" valvular heart disease and treatment with pergolide (3): in several cases, the valvulopathy improved when pergolide was discontinued (4). Valvular heart damage has also been reported with the ergot-derived dopamine agonists bromocriptine and cabergoline (5,6).

Two recent studies (7,8) have further demonstrated that both pergolide and cabergoline are associated with an increased risk of new cardiac valve regurgitation in patients treated for Parkinson's disease.

The valvular abnormalities seen with ergot-derived dopamine agonists are similar to those observed in patients receiving ergot alkaloid agents (such as ergotamine and methysergide) in the treatment of migraine, or fenfluramine and dexfenfluramine in the treatment of obesity. These abnormalities also closely resemble carcinoid-related valvulopathies (9).

Cardiac valve disease has never been reported in patients with prolactinomas who require treatment with dopamine-agonists even life-long (1). At variance with patients with Parkinson's disease, patients with prolactinomas are younger and are treated with an average dose of dopamine-agonists that is significantly lower (median bromocriptine dose 5 mg/day and median cabergoline dose 1 mg/week). Because of the young age of treatment beginning (most patients with microprolactinomas start dopamine-agonist treatment in early adulthood), treatment might be continued for over 3 decades: the cumulative risk of low doses of dopamine agonists for such a long period of treatment is currently unknown.

To assess the prevalence of cardiac valve disease in patients treated with cabergoline, we wish to perform an echocardiography screening in a large representative sample of patients with prolactinoma who were treated with cabergoline for at least 12 months and in a group of control subjects recruited prospectively. We wish to evaluate the severity of regurgitation for the mitral, aortic, and tricuspid valves. Changes in cardiac valve apparatus was compared with treatment duration and cumulative cabergoline dose.

DETAILED DESCRIPTION:
Within one week from a clinical observation in the outpatient service, all patients will be admitted to the hospital for a complete endocrine screening, a cardiological visit that will include an electrocardiogram and an echocardiogram.

The endocrine profile will include measurement of IGF-I, PRL, FSH, LH, 17-β-estradiol, testosterone, FT3, FT4, TSH, and cortisol at 8.00 in the morning after an overnight fasting.

The clinical profile will include blood pressure measurement at the right arm, with the subjects in relaxed sitting position. The average of six measurements (three taken by each of two examiners, in the same day of echocardiography, between 8.00-9.00 in the morning) with a mercury sphygmomanometer will be used in all analysis. According with the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (10), hypertension, if present, is classified as mild (Stage 1) when the SBP or DBP were between 140 and 159 mmHg and between 90 and 99 mmHg, respectively; severe (Stage 2) when the SBP or DBP were >160 and >100 mmHg respectively; pre-hypertension is defined as SBP >120¬ and <140 and DBP >80 and <90 mmHg. Heart rate will be also measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented hyperprolactinemia receiving continuous treatment with cabergoline only for at least 12 months
* Newly diagnosed patients with prolactinoma never previously receiving dopamine agonists treatment

Exclusion Criteria:

* A history of cardiac valve abnormalities,
* Previous use of anorectic drugs or other ergot-derived drugs,
* Treatment with cabergoline for less than 12 months,
* Valve calcification, valve regurgitation associated with annular dilatation or excessive leaflet motion,
* Mitral regurgitation associated with left ventricular wall-motion abnormalities or left ventricular dilatation,
* Withdrawal from cabergoline treatment for longer than 1 month, according with our treatment protocol (11).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three different study populations will be studied.
  * Group 1) Patients already receiving treatment with cabergoline for at least 12 months
  * Group 2) Newly diagnosed patients with hyperprolactinemia who never received treatment with dopamine-agonists
  * Group 3) Non hyperprolactinemic subjects matched with the patients for sex and age to be used as controls.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of regurgitation (graded as mild, moderate, severe) at any cardiac valve. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria AL Colao, Prof., Principal Investigator — Federico II University
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, University Federico II of Naples, Via S. Pansini 5 Naples, Italy

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Result] Gillam MP, Molitch ME, Lombardi G, Colao A. Advances in the treatment of prolactinomas. Endocr Rev. 2006 Aug;27(5):485-534. doi: 10.1210/er.2005-9998. Epub 2006 May 26. PMID 16705142
- [Result] Nutt JG, Wooten GF. Clinical practice. Diagnosis and initial management of Parkinson's disease. N Engl J Med. 2005 Sep 8;353(10):1021-7. doi: 10.1056/NEJMcp043908. No abstract available. PMID 16148287
- [Result] Flowers CM, Racoosin JA, Lu SL, Beitz JG. The US Food and Drug Administration's registry of patients with pergolide-associated valvular heart disease. Mayo Clin Proc. 2003 Jun;78(6):730-1. doi: 10.4065/78.6.730. No abstract available. PMID 12934784
- [Result] Van Camp G, Flamez A, Cosyns B, Weytjens C, Muyldermans L, Van Zandijcke M, De Sutter J, Santens P, Decoodt P, Moerman C, Schoors D. Treatment of Parkinson's disease with pergolide and relation to restrictive valvular heart disease. Lancet. 2004 Apr 10;363(9416):1179-83. doi: 10.1016/S0140-6736(04)15945-X. PMID 15081648
- [Result] Pinero A, Marcos-Alberca P, Fortes J. Cabergoline-related severe restrictive mitral regurgitation. N Engl J Med. 2005 Nov 3;353(18):1976-7. doi: 10.1056/NEJM200511033531822. No abstract available. PMID 16267335
- [Result] Serratrice J, Disdier P, Habib G, Viallet F, Weiller PJ. Fibrotic valvular heart disease subsequent to bromocriptine treatment. Cardiol Rev. 2002 Nov-Dec;10(6):334-6. doi: 10.1097/00045415-200211000-00005. PMID 12390688
- [Result] Schade R, Andersohn F, Suissa S, Haverkamp W, Garbe E. Dopamine agonists and the risk of cardiac-valve regurgitation. N Engl J Med. 2007 Jan 4;356(1):29-38. doi: 10.1056/NEJMoa062222. PMID 17202453
- [Result] Zanettini R, Antonini A, Gatto G, Gentile R, Tesei S, Pezzoli G. Valvular heart disease and the use of dopamine agonists for Parkinson's disease. N Engl J Med. 2007 Jan 4;356(1):39-46. doi: 10.1056/NEJMoa054830. PMID 17202454
- [Result] Botero M, Fuchs R, Paulus DA, Lind DS. Carcinoid heart disease: a case report and literature review. J Clin Anesth. 2002 Feb;14(1):57-63. doi: 10.1016/s0952-8180(01)00353-1. PMID 11880025
- [Result] Colao A, Di Sarno A, Cappabianca P, Di Somma C, Pivonello R, Lombardi G. Withdrawal of long-term cabergoline therapy for tumoral and nontumoral hyperprolactinemia. N Engl J Med. 2003 Nov 20;349(21):2023-33. doi: 10.1056/NEJMoa022657. PMID 14627787
- [Derived] Auriemma RS, Pivonello R, Perone Y, Grasso LF, Ferreri L, Simeoli C, Iacuaniello D, Gasperi M, Colao A. Safety of long-term treatment with cabergoline on cardiac valve disease in patients with prolactinomas. Eur J Endocrinol. 2013 Aug 28;169(3):359-66. doi: 10.1530/EJE-13-0231. Print 2013 Sep. PMID 23824978
- [Derived] Colao A, Galderisi M, Di Sarno A, Pardo M, Gaccione M, D'Andrea M, Guerra E, Pivonello R, Lerro G, Lombardi G. Increased prevalence of tricuspid regurgitation in patients with prolactinomas chronically treated with cabergoline. J Clin Endocrinol Metab. 2008 Oct;93(10):3777-84. doi: 10.1210/jc.2007-1403. Epub 2008 Aug 5. PMID 18682513